CLINICAL TRIAL: NCT06152861
Title: Multicenter, Randomized, Double-Masked, Active-Controlled, Parallel Group Phase 2 Trial Evaluating the Safety and Efficacy of Travoprost Ophthalmic Topical Cream in Subjects With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Travoprost Ophthalmic Topical Cream for Open-angle Glaucoma or Ocular Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLK-311-01
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Travoprost Ophthalmic Topical Cream low-dose (Experimental): Travoprost Ophthalmic Topical Cream low-dose administered once-daily in the evening for 28 days
  Interventions: Drug: Travoprost Ophthalmic Topical Cream low-dose
- Travoprost Ophthalmic Topical Cream mid-dose (Experimental): Travoprost Ophthalmic Topical Cream mid-dose administered once-daily in the evening for 28 days
  Interventions: Drug: Travoprost Ophthalmic Topical Cream mid-dose
- Travoprost Ophthalmic Topical Cream high-dose (Experimental): Travoprost Ophthalmic Topical Cream high-dose administered once-daily in the evening for 28 days
  Interventions: Drug: Travoprost Ophthalmic Topical Cream high-dose
- Timolol maleate ophthalmic solution, 0.5% (Active Comparator): Timolol maleate ophthalmic solution, 0.5% administered twice daily, morning and evening, for 28 days
  Interventions: Drug: Timolol maleate ophthalmic solution, 0.5%
- Travoprost ophthalmic solution, 0.004% (Active Comparator): Travoprost ophthalmic solution, 0.004% administered once daily in the evening for 28 days
  Interventions: Drug: Travoprost Ophthalmic Solution, 0.004%

INTERVENTIONS:
Drug: Travoprost Ophthalmic Topical Cream low-dose — travoprost ophthalmic topical cream low-dose once daily in the evening to both eyes
  Arms: Travoprost Ophthalmic Topical Cream low-dose
Drug: Travoprost Ophthalmic Topical Cream mid-dose — travoprost ophthalmic topical cream mid-dose once daily in the evening to both eyes
  Arms: Travoprost Ophthalmic Topical Cream mid-dose
Drug: Travoprost Ophthalmic Topical Cream high-dose — travoprost ophthalmic topical cream high-dose once daily in the evening to both eyes
  Arms: Travoprost Ophthalmic Topical Cream high-dose
Drug: Timolol maleate ophthalmic solution, 0.5% — timolol maleate ophthalmic solution, 0.5% twice daily (morning & evening) to both eyes
  Arms: Timolol maleate ophthalmic solution, 0.5%
Drug: Travoprost Ophthalmic Solution, 0.004% — travoprost ophthalmic solution, 0.004% once daily in the evening to both eyes
  Arms: Travoprost ophthalmic solution, 0.004%

SUMMARY:
The goal of this clinical trial is to learn about the safety of Travoprost Ophthalmic Topical Cream and how well it works in lowering high intraocular pressure (IOP) in patients with open-angle glaucoma (OAG) or ocular hypertension (OHT).

A low dose, medium dose and high dose of Travoprost Ophthalmic Topical Cream will be compared to timolol maleate ophthalmic solution, 0.5% and to travoprost ophthalmic solution, 0.004%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older at the Screening Visit;
* Willing and able to provide written informed consent on the IRB/IEC-approved informed consent form;
* Diagnosis of OAG (including pigmentary and pseudoexfoliative) or OHT in both eyes;
* Qualifying IOP in the study eye;
* Best-corrected visual acuity of approximately 20/80 Snellen in each eye

Exclusion Criteria:

* Sensitivity or allergy to travoprost or timolol;
* Bronchial asthma, a history of bronchial asthma, or severe chronic obstructive pulmonary disease;
* History of or current sinus bradycardia, second- or third-degree atrioventricular block, overt cardiac failure, or cardiogenic shock;
* History of cerebrovascular insufficiency;
* Any form of glaucoma other than open-angle glaucoma
* Advanced visual field loss or cup-to-disc ratio of 0.8 or greater
* Non-qualifying prior surgeries or procedures in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
change from baseline in mean diurnal IOP in the study eye | Day 29
  Day 29 mean diurnal IOP minus Baseline mean diurnal IOP in the study eye

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Glaukos Corporation
Locations (1):
- Glaukos Clinical Study Site, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No